CLINICAL TRIAL: NCT07383558
Title: Does Targeting the Sural Nerve in Addition to the Posterior Tibial Nerve Increase the Effectiveness of Pulsed Radiofrequency Treatment in Chronic Plantar Heel Pain?
Brief Title: Effect of Additional Sural Nerve PRF in Chronic Heel Pain
Status: Recruiting | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Supervisor Investigator, Diskapi Teaching and Research Hospital
Other Study IDs: Sural-Posterior Tibial PRF
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Chronic Plantar Heel Pain; Plantar Fasciitis; Spur, Heel
Keywords: posterior tibial nerve, sural nerve, chronic heel pain, plantar heel pain
MeSH Terms: conditions — Fasciitis, Plantar; Heel Spur | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Posterior tibial nerve PRF: Patients with chronic plantar heel pain who received ultrasound-guided pulsed radiofrequency treatment applied only to the posterior tibial nerve as part of routine clinical care.
  Interventions: Procedure: Pulsed radiofrequency
- Posterior tibial + sural nerve PRF: Patients with chronic plantar heel pain who received ultrasound-guided pulsed radiofrequency treatment applied to both the posterior tibial nerve and the sural nerve as part of routine clinical care.
  Interventions: Procedure: Pulsed radiofrequency

INTERVENTIONS:
Procedure: Pulsed radiofrequency — Ultrasound-guided pulsed radiofrequency applied to the posterior tibial nerve, with or without additional application to the sural nerve.

SUMMARY:
This observational study aims to compare the effectiveness of pulsed radiofrequency (PRF) treatment applied to the posterior tibial nerve alone versus PRF applied to both the posterior tibial and sural nerves in patients with chronic plantar heel pain. Outcomes will be assessed using the Visual Analog Scale (VAS) and the American Orthopaedic Foot and Ankle Society (AOFAS) hindfoot score at baseline, 1 month, and 3 months after treatment.

DETAILED DESCRIPTION:
Chronic plantar heel pain is a common condition frequently managed with interventional pain procedures. In routine clinical practice, pulsed radiofrequency (PRF) is commonly applied to the posterior tibial nerve under ultrasound guidance. In selected patients, PRF is additionally applied to the sural nerve based on clinical judgment.

This observational study includes patients who have already undergone PRF treatment as part of standard care in the Algology Clinic. Patients will not be randomized, and no modification to treatment plans will be made for study purposes. Patients will be divided into two groups: those who received PRF to the posterior tibial nerve alone, and those who received PRF to both the posterior tibial and sural nerves. Pain intensity and functional outcomes will be retrospectively evaluated and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 65 years

Presence of chronic plantar heel pain

Baseline VAS score >5

Exclusion Criteria:

History of foot fracture or tumor

Pregnancy

Coagulopathy or use of antiplatelet therapy

Cognitive impairment preventing informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 65 years with chronic plantar heel pain who underwent ultrasound-guided pulsed radiofrequency (PRF) treatment of the posterior tibial nerve, with or without additional PRF of the sural nerve, as part of routine clinical care in the Algology Clinic. Patients were included if they had a baseline Visual Analog Scale (VAS) pain score greater than 5. All treatments were completed prior to study enrollment, and no changes were made to clinical management for research purposes.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
VAS | Baseline, 1 month, and 3 months post-procedure
  Change in pain intensity assessed by Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
AOFAS | Baseline, 1 month, and 3 months post-procedure
  Functional improvement assessed by American Orthopaedic Foot and Ankle Society (AOFAS) Hindfoot Score

CONTACTS AND LOCATIONS:
Locations (1):
- Ayse Betul Acar, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No